CLINICAL TRIAL: NCT00624078
Title: Treatment Protocol for Use of Anascorp™ in Patients With Scorpion Sting Envenomation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto Bioclon S.A. de C.V. (Industry)
Collaborators: University of Arizona (Other)
Responsible Party: Walter Garcia U. MD/Clinical Research Manager, Instituto Bioclon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL-03/07
Record Dates: First submitted 2007-12-26; First posted 2008-02-26 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Scorpion Sting Envenomation
Keywords: faboterapics; treatment; scorpion sting; envenomation
MeSH Terms: conditions — Scorpion Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients who arrive to emergency room with scorpion sting envenomation will be evaluated according to inclusion/exclusion criteria. After informed consent has been signed they will be assigned to unique treatment arm with Anascorp.
  Interventions: Drug: Antivenin Centruroides (scorpion) F(ab)2 Anascorp™

INTERVENTIONS:
Drug: Antivenin Centruroides (scorpion) F(ab)2 Anascorp™ — three vials diluted in 20 to 50 mL normal saline administered intravenously. Subsequent single vial doses of Anascorp, up to a total of five vials administered at thirty minutes intervals until resolution of symptoms.

SUMMARY:
This treatment protocol will enable therapeutic use of Anascorp in the management of systemic manifestations of scorpion sting envenomation, in patients for whom antivenom would otherwise be unavailable. The working hypotheses are as follows:

1. The investigational antivenom is safe as treatment of scorpion sting envenomation.
2. The investigational antivenom is effective as treatment of scorpion sting envenomation.

DETAILED DESCRIPTION:
The purpose of this Open Label, Multi-Center Treatment Protocol, phase III trial is to examine the safety and efficacy of Anascorp, for treatment of patients envenomed by scorpion sting.

The treatment protocol, including up to 25 Arizona sites, increases the total number of subjects receiving Anascorp™, and can provide supplemental safety data for the review process. At the same time, it will prevent a public health crisis in rural Arizona by replacing the dwindling supply of local antivenom before an BLA is approved.

Patients who arrive at the emergency clinic presenting with scorpion sting symptoms will be evaluated for treatment with Anascorp.

Each patient who qualifies for entry into the study, according to inclusion/exclusion criteria, is assigned a patient number in sequential order of entry. Approximately 100 patients could be enrolled in the study per year.

After informed consent has been obtained, a baseline history and physical will be obtained and documented in the patient's chart. This will include an evaluation of the symptoms of systemic scorpion envenomation. The patient's vital signs (blood pressure, pulse and respiration) will be taken. The patient will be questioned as to concomitant medications. Demographic data will also be collected.

Three vials of Anascorp will be administered in a total volume of 50 mL, intravenous over not less than 10 minutes or as permitted by IV access. If clinically indicated by systemic signs, a second dose (one vial) will be administered if clinically indicated by systemic signs. One additional dose may be administered 30 minutes later if indicated by clinically significant signs of envenomation. When clinically significant signs have been absent for at least 30 minutes, a final physical assessment will take place and the patient will be discharged to home.

Twenty four hours and fourteen days after Anascorp™ treatment, all patients will be monitored for signs and symptoms of adverse events, including acute hypersensitivity reactions (anaphylactic and/or anaphylactoid reactions) and delayed serum sickness. All patients who received study drug will be included in the final analyses.

For the individual patient, the study starts at the time the consent is signed and ends at the 14 day telephone interview. The outcome is assessed 14 days after discharge by telephone interview.

Concomitant therapy and medications may be used at any time as needed. All concomitant medication must be documented in the CRF from time of entry into the study until the 14 day follow up telephone interview..

ELIGIBILITY:
Inclusion Criteria:

* Males and females of any age presenting for emergency treatment with clinically important systemic signs of scorpion sting envenomation
* Signed written Informed Consent by patient or legal guardian

Exclusion Criteria:

* Allergy to horse serum

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1426 (Actual)
Dates: Start 2005-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the adverse events profile of each patient | immediately after treatment, 24 hrs and 14 days.

SECONDARY OUTCOMES:
Resolution of systemic signs of scorpion envenomation | after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Boyer, M.D, Principal Investigator — VIPER Institute; Walter Garcia, M.D, Study Chair — Instituto Bioclon S.A. de C.V.
Locations (18):
- United States (18):
  - Casa Grande Regional Medical Center, Casa Grande, Arizona
  - Chandler Regional, Chandler, Arizona
  - Southeast Arizona Medical Center, Douglas, Arizona
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Banner Thunderbird Medical Center, Glendale, Arizona
  - Banner Baywood Medical Center, Mesa, Arizona
  - Gila Health Resources, Morenci, Arizona
  - Holy Cross Hospital, Nogales, Arizona
  - Maricopa Medical Center, Phoenix, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - John C. Lincoln, Phoenix, Arizona
  - Mt. Graham Regional Medical Center, Safford, Arizona
  - San Carlos Indian Hospital, San Carlos, Arizona
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - University Medical Center, Tucson, Arizona
  - St. Mary's Hospital, Tucson, Arizona
  - Whiteriver IHS Hospital, Whiteriver, Arizona

REFERENCES:
- [Background] Vazquez H, Chavez-Haro A, Garcia-Ubbelohde W, Mancilla-Nava R, Paniagua-Solis J, Alagon A, Sevcik C. Pharmacokinetics of a F(ab')2 scorpion antivenom in healthy human volunteers. Toxicon. 2005 Dec 1;46(7):797-805. doi: 10.1016/j.toxicon.2005.08.010. Epub 2005 Sep 28. PMID 16197974
- [Background] Likes K, Banner W Jr, Chavez M. Centruroides exilicauda envenomation in Arizona. West J Med. 1984 Nov;141(5):634-7. PMID 6516334
- [Background] Lai MW, Klein-Schwartz W, Rodgers GC, Abrams JY, Haber DA, Bronstein AC, Wruk KM. 2005 Annual Report of the American Association of Poison Control Centers' national poisoning and exposure database. Clin Toxicol (Phila). 2006;44(6-7):803-932. doi: 10.1080/15563650600907165. PMID 17015284
- [Background] Gibly R, Williams M, Walter FG, McNally J, Conroy C, Berg RA. Continuous intravenous midazolam infusion for Centruroides exilicauda scorpion envenomation. Ann Emerg Med. 1999 Nov;34(5):620-5. doi: 10.1016/s0196-0644(99)70164-2. PMID 10533010
- [Background] Riley BD, LoVecchio F, Pizon AF. Lack of scorpion antivenom leads to increased pediatric ICU admissions. Ann Emerg Med. 2006 Apr;47(4):398-9. doi: 10.1016/j.annemergmed.2005.11.042. No abstract available. PMID 16546632